CLINICAL TRIAL: NCT04177966
Title: The Effect of Pre-operative Videotape Before a Planned Cesarean Section on Anxiety Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Eyal Rom, MD, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMC-19-130
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Cesarean Section Complications; Pain, Postoperative; Analgesia
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Women will be recruited for research at the time of admission preoperatively According to randomization women will be divided into two groups - intervention and control
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women watching the pre-prepared video before surgery (Experimental): Women undergoing primary elective cesarean surgery at term The day before surgery the women will watch a pre-prepared video, approximately 10 minutes in length, showing in detail the course of events around the operation
  Interventions: Behavioral: pre-prepared video describing the cesarean surgery
- women not watching the pre-prepared video before surgery (Placebo Comparator): Women undergoing primary elective cesarean surgery at term Women will receive general information about the surgery as part of informed consent, without watching a pre- prepared film.
  Interventions: Behavioral: general information

INTERVENTIONS:
Behavioral: pre-prepared video describing the cesarean surgery — a pre-prepared video, approximately 10 minutes in length, showing in detail the course of events around the operation - from the woman's perspective - from the time they were admitted to the department, preparation for surgery, entrance to the operating r
  Arms: women watching the pre-prepared video before surgery
Behavioral: general information — In the control group - women will receive general information about the surgery as part of informed consent, without watching a pre-prepared film.
  Arms: women not watching the pre-prepared video before surgery

SUMMARY:
The study aim is to examine the relationship between providing information to women prior to elective cesarean delivery and anxiety levels around surgery.

the patients will be assigned into two groups - intervention and control. In the intervention group - the day before surgery the women will watch a pre-prepared video showing in detail the course of events around the operation.

the level of anxiety, pain level and Intake of Analgesics will be compared between the two groups

DETAILED DESCRIPTION:
Women will be recruited for research at the time of admission preoperatively. According to randomization women will be divided into two groups - intervention and control In the intervention group - the day before surgery the women will watch a pre-prepared video, approximately 10 minutes in length, showing in detail the course of events around the operation - from the woman's perspective - from the time they were admitted to the department, preparation for surgery, entrance to the operating room, anesthesia procedure, surgery Itself, post-operative recovery and recovery course in maternity ward.

The movie will be shown to the patient by one of the study investigators. In the control group - women will receive general information about the surgery as part of the routine informed consent process, without watching a pre- prepared film.

the level of anxiety, pain level and Intake of Analgesics will be compared between the two groups

ELIGIBILITY:
Inclusion Criteria:

* First cesarean surgery

Exclusion Criteria:

* Women who have had surgery beyond age 2 years
* Women with anxiety disorders
* Women with comorbidity that might alter cortisol and catecholamine excretion,
* Women with comorbidity associated with severe pain that might distort pain ratings
* Women with psychiatric comorbidity that might reduce the ability to understand the videotape and questionnaires
* Women who consume any medication that might affect urinary excretion of cortisol
* Women undergoing cesarean surgery due to obstetric complication (gestational hypertension, pre-eclampsia, gestational diabetes mellitus)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in anxiety level between the two groups at one hour before surgery. | 3 points: before watching the movie (t1), one hour before surgery (t2), 8 hours after the surgery (t3).
  To assess a patient's anxiety response to a given situation, the investigators will use State Trait Anxiety Scale (STAI) questionnaire. The questionnaire consists of two sets of 20 different questions that can be answered from 1 to 4. The first (state subscale) assesses a current anxiety condition, while the second (trait subscale) assesses personality characteristics.
  This questionnaire was found to be valid for use in a study of a pregnant women population. High scores indicate high levels of anxiety Although the outcome is the The difference in anxiety level between the two groups at one hour before surgery, the investigators will assess the baseline anxiety level and 8 hours after the surgery, for inter-group comparison.

SECONDARY OUTCOMES:
Maternal complications | during the time of hospitalization after delivery, up to 1 month
  any obstetrical complication
Change from baseline biochemical anxiety level at 6 hours interval following the surgery | 2 points: the morning before surgery (c1) and 6 hours following the surgery (c2)
  Cortisol blood levels taken 6 hours following the surgery. Although the outcome is the change from baseline level at 6 hours following the surgery, the investigators will assess the cortisol level 6 hours after the surgery for inter-group comparison.
Change from baseline pain level at 8 hours after surgery | 3 points: before watching the movie (t1), one hour before the surgery (t2), 8 hours after the surgery (t3).
  To assess a patient's pain level, the investigators will use visual analog scale (VAS)- scale for patient self-reporting of pain. 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-10 represents severe pain). a lower pain level 8 hours after surgery is a better outcome Although the outcome is the change from baseline level at 8 hours after the surgery, the investigators will assess the pain level before the surgery for inter-group comparison.

CONTACTS AND LOCATIONS:
Overall Officials: eyal rom, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Haemek Medical Center, Afula, Israel